CLINICAL TRIAL: NCT01061931
Title: HD Mesh Ablator Versus Cryoballoon Pulmonary Vein Ablation of Symptomatic Paroxysmal Atrial Fibrillation - Efficiency and Safety of PV Ablation Systems
Brief Title: Mesh Ablator Versus Cryoballoon Pulmonary Vein Ablation of Symptomatic Paroxysmal Atrial Fibrillation
Acronym: MACPAF
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: reason
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Jochen B. Fiebach, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MACPAF; 4-087-08 (Other: ethic's committee Charité Berlin)
Record Dates: First submitted 2010-02-02; First posted 2010-02-03 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Symptomatic Paroxysmal Atrial Fibrillation
Keywords: MRI; left-sided atrial catheter ablation; paroxysmal atrial fibrillation; cryoballoon technique; mesh ablator catheter; stroke; silent stroke; major complications
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arctic Front® catheter (Active Comparator)
  Interventions: Procedure: Arctic Front® catheter vs. HD Mesh Ablator® catheter
- HD Mesh Ablator® catheter (Active Comparator)
  Interventions: Procedure: Arctic Front® catheter vs. HD Mesh Ablator® catheter

INTERVENTIONS:
Procedure: Arctic Front® catheter vs. HD Mesh Ablator® catheter — Pulmonary vein ablation in patients with symptomatic paroxysmal atrial fibrillation using the Arctic Front® catheter versus the HD Mesh Ablator® catheter

SUMMARY:
The purpose of this prospective randomized single-center trial is to compare efficiency and safety of two pulmonary vein ablation systems in patients with symptomatic paroxysmal atrial fibrillation using the Arctic Front® versus the HD Mesh Ablator® catheter.

DETAILED DESCRIPTION:
Primary objective:

• Efficacy of pulmonary vein isolation defined by achieving an exit block for all pulmonary veins per patient.

Secondary objectives:

* Detecting (silent) cerebral thromboembolism using neuro(psychological) tests and brain MRI prior and within 2 days after PV ablation.
* Detecting (silent) cerebral thromboembolism using neuro(psychological) tests and brain MRI within 6 months after PV ablation.
* Determination of spontaneous recurrence rate of atrial fibrillation using a subcutaneously implanted loop recorder (Reveal XT®).
* Characterization of non-neurological major complications (death, atrial-esophageal fistula, pulmonary vein stenosis, pericardial tamponade)
* Rate of iatrogenic interatrial septal defects after transseptal puncture for PV ablation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ECG-documented symptomatic paroxysmal atrial fibrillation and at least one ineffective antiarrhythmic drug treatment

Exclusion Criteria:

* Previous ablation procedure for atrial fibrillation or cardiac surgery within 3 months
* Left atrial diameter > 50mm or ejection fraction < 35%
* Instable coronary artery disease or clinically relevant cardiac valve insufficiency
* Hyperthyroidism, pregnancy or lactation; coumadin or heparin intolerance
* Concomitant disease with expected lifespan < 2 years
* Contraindications for MRI or acute cerebral infarction detected by brain MRI immediately (< 24 hours) before catheter ablation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Efficacy of pulmonary vein isolation defined by achieving an exit block for all pulmonary veins per patient | During ablation procedure

SECONDARY OUTCOMES:
Detecting (silent) cerebral thromboembolism using neuro(psychological) tests and brain MRI | within 2 days after catheter ablation
Detecting (silent) cerebral thromboembolism using neuro(psychological) tests and brain MRI | 6 months after catheter ablation
Determination of spontaneous recurrence rate of atrial fibrillation using a subcutaneously implanted loop recorder (Reveal XT®) | 1 year after catheter ablation
Characterization of non-neurologic major complications (death, atrial-esophageal fistula, pulmonary vein stenosis, pericardial tamponade) | within 1 month after catheter ablation
Rate of iatrogenic interatrial septal defects after transseptal puncture for left-sided atrial catheter ablation | 1 year after catheter ablation

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Schirdewan, MD, Principal Investigator — Department of Cardiology, Charité - University Medicine Berlin, Germany.; Jochen B Fiebach, MD, Principal Investigator — Center for Stroke Research Berlin
Locations (1):
- Charité, University Medicine Berlin, Campus Benjamin Franklin, Hindenburgdamm 30, Berlin, Germany

REFERENCES:
- [Derived] Herm J, Schirdewan A, Koch L, Wutzler A, Fiebach JB, Endres M, Kopp UA, Haeusler KG. Impact of atrial fibrillation burden on cognitive function after left atrial ablation - Results of the MACPAF study. J Clin Neurosci. 2020 Mar;73:168-172. doi: 10.1016/j.jocn.2019.12.030. Epub 2020 Jan 25. PMID 31992513
- [Derived] Schirdewan A, Herm J, Roser M, Landmesser U, Endres M, Koch L, Haeusler KG. Loop Recorder Detected High Rate of Atrial Fibrillation Recurrence after a Single Balloon- or Basket-Based Ablation of Paroxysmal Atrial Fibrillation: Results of the MACPAF Study. Front Cardiovasc Med. 2017 Feb 13;4:4. doi: 10.3389/fcvm.2017.00004. eCollection 2017. PMID 28243592
- [Derived] Herm J, Fiebach JB, Koch L, Kopp UA, Kunze C, Wollboldt C, Brunecker P, Schultheiss HP, Schirdewan A, Endres M, Haeusler KG. Neuropsychological effects of MRI-detected brain lesions after left atrial catheter ablation for atrial fibrillation: long-term results of the MACPAF study. Circ Arrhythm Electrophysiol. 2013 Oct;6(5):843-50. doi: 10.1161/CIRCEP.113.000174. Epub 2013 Aug 29. PMID 23989301
- [Derived] Haeusler KG, Koch L, Herm J, Kopp UA, Heuschmann PU, Endres M, Schultheiss HP, Schirdewan A, Fiebach JB. 3 Tesla MRI-detected brain lesions after pulmonary vein isolation for atrial fibrillation: results of the MACPAF study. J Cardiovasc Electrophysiol. 2013 Jan;24(1):14-21. doi: 10.1111/j.1540-8167.2012.02420.x. Epub 2012 Aug 22. PMID 22913568
- [Derived] Koch L, Haeusler KG, Herm J, Safak E, Fischer R, Malzahn U, Werncke T, Heuschmann PU, Endres M, Fiebach JB, Schultheiss HP, Schirdewan A. Mesh ablator vs. cryoballoon pulmonary vein ablation of symptomatic paroxysmal atrial fibrillation: results of the MACPAF study. Europace. 2012 Oct;14(10):1441-9. doi: 10.1093/europace/eus084. Epub 2012 Apr 20. PMID 22523379
- [Derived] Haeusler KG, Koch L, Ueberreiter J, Coban N, Safak E, Kunze C, Villringer K, Endres M, Schultheiss HP, Fiebach JB, Schirdewan A. Safety and reliability of the insertable Reveal XT recorder in patients undergoing 3 Tesla brain magnetic resonance imaging. Heart Rhythm. 2011 Mar;8(3):373-6. doi: 10.1016/j.hrthm.2010.11.008. Epub 2010 Nov 9. PMID 21070885
- [Derived] Haeusler KG, Koch L, Ueberreiter J, Endres M, Schultheiss HP, Heuschmann PU, Schirdewan A, Fiebach JB. Stroke risk associated with balloon based catheter ablation for atrial fibrillation: Rationale and design of the MACPAF Study. BMC Neurol. 2010 Jul 21;10:63. doi: 10.1186/1471-2377-10-63. PMID 20663131